CLINICAL TRIAL: NCT01883115
Title: A Prospective Study Comparing Telescopic vs. Balloon Dissection in Single Incision Laparoscopic Inguinal Herniorraphy (SILTELESCOPIC)
Acronym: SILTelescopic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Sydney Hernia Specialists Clinic (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Dr Hanh Minh Tran, Director, The Sydney Hernia Specialists Clinic
Other Study IDs: SILTelescopic
Record Dates: First submitted 2013-06-16; First posted 2013-06-21 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Inguinal Hernia
Keywords: Telescopic extraperitoneal dissection; Single incision laparosocpic surgery; Inguinal hernia; Triport system
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Telescopic group: All eligible patients referred with inguinal/femoral hernias will be enrolled into the study from February 2013

SUMMARY:
Our recent prospective randomized controlled study comparing single-port vs. multiport laparoscopic total extraperitoneal inguinal herniorraphy (NCT 01660048) demonstrated superiority of the single-port technique in reducing post-op pain/analgesic requirements, quicker return to work/normal physical activities and improved cosmetic scar scores. During this study all patients underwent the initial extraperitoneal dissection with the distension balloon. However, the balloon itself costs AU $380 per device which represents a significant percentage of the overall cost of the procedure (when the hospital/operating rooms cost is approximately AU $2500 for a unilateral laparoscopic inguinal hernia repair) especially if only unilateral inguinal herniorraphy is performed.

The European Hernia Society Guidelines encourage the use of the distension balloon for the initial distension/dissection of the extraperitoneal space especially during the learning curve. This recommendation arises from the fact that during the conventional multiport repair the umbilical port allows only the insertion of the laparoscope and the extraperitoneal space cannot easily be dissected with the scope itself, especially in patients with well-developed linea alba extending down to the pubic symphysis, and the camera itself, if used as dissection device, would become smudged and it would have to be repeatedly withdrawn for cleaning. Yet this must occur since the extraperitoneal space must be dissected in the midline sufficiently for safe insertion of two additional 5 mm ports for insertion of dissecting instruments in order to complete the extraperitoneal space dissection and the repair.

With single incision laparoscopic surgery the use of the Triport™ system ensure that the port can be place under direct vision into the extraperitoneal space when the scope and two dissecting instruments can be safely inserted at the outset. In this way the extraperitoneal space can be dissected under direct vision. The balloon dissection is essentially a blind dissection even though the balloon distension is being observed by the scope, incorrect tissue planes can be entered ie the dissection can occur below the pre-peritoneal fascia exposing the nerves in the groin with the potential risks for nerve damage and entrapment. This is an argument that surgeons who practise transabdominal preperitoneal inguinal hernia repair use to justify their superior technique over the TEP repair because, in the TAPP repair, the peritoneum is carefully dissected free from and leaving the underlying preperitoneal fascia intact.

While the use of the balloon, when some 25 "pumps" of air are used during the insufflation, to create a significant space to place not only the two 5 mm ports but also to create a significant extraperitoneal dissection when usually only the lateral space and the hernia sac need to be dissected this is not always possible. In patients who have had previous lower abdominal surgery including previous anterior inguinal herniorraphy (especially if the mesh plug is used) the balloon dissention is normally judicious as one cannot predict whether there are any significant peritoneal or even bowel adhesions. Consequently, in such cases, the balloon distension is normally confined to an area just inferior to the umbilical port and superior to the pubic symphysis so that there is just enough extraperitoneal dissection to place the two 5 mm trocars. Usually this means only using only 5 pumps of air in the distension balloon for placement of two 5 mm trocars. Then the dissection of the extraperitonealy space under direct vision can take place. The use of the distension balloon in such cases represents an enormous waste of resources since AU $380 is spent just to create enough space to place the two 5 mm ports and hence allowing the insertion of the dissecting instruments. With the Triport+™ port the dissecting instruments can easily be placed in the extraperitoneal space and the dissection can begin under direct vision hence achieving the same safe dissection that TAPP surgeons claim to perform.

In this study we aim to look at the safety and efficacy of telescopic vs. balloon dissection by prospectively comparing a similar former group of patients to the ones who had previously undergone single-port inguinal herniorraphy with balloon dissection in our previous study (NCT 01660048).

All patients having surgical treatment of groin hernia at St Luke's and Holroyd Private Hospitals are subject to very careful assessment and study. All patients are requested to report immediately if there are any problems.

DETAILED DESCRIPTION:
This study will compare the extraperitoneal dissection during single-port laparoscopic total extraperitoneal repair of inguinal/femoral hernias using the traditional balloon dissection and the telescopic dissection techniques.

Laparoscopic hernia repair was first introduced in 1990. The uptake rate was slow to start off with such that in 1994 only 9.7% of all inguinal hernias were performed laparoscopically However, in 2012, the figure now stands at 48% Australia-wide. (www.medicareaustralia.gov.au). Indeed, in the State of New South Wales this figure stands at 51%, which means that it is the commonest operation performed for inguinal hernias in this State.

Up to 2009, the laparoscopic hernia repair involves the insertion of 3 ports: 10mm port in the infra-umbilical region for the camera via a 2 cm incision and 2 x 5 mm working ports usually in the midline for the dissecting instruments via 2 x 10 mm incisions. These ports are called secondary trocars which are usually sharp. Their insertion has the potential to cause bowel and vascular injuries.

The European Hernia Society guidelines (www.herniaweb.org) on the treatment of inguinal hernias have shown (conventional) endoscopic techniques to be associated with higher rates of port-site hernias and visceral injuries especially during the learning curve period.

A recent study of 37,000 gynaecological laparoscopies in the US showed a bowel injury rate of 0.16%; a third of these led to the death of the patients. 22% of all bowel injuries resulted from the insertion of secondary trocars (www.danaise.com/vascular_and_bowel_injuries_duri.htm).

Another report from a large hernia centre in the US showed that in the first 300 transabdominal preperitoneal (TAPP) repairs 2 bowel injuries (and one bladder injury) were observed. Indeed, when these investigators changed the technique to a TEP repair they also observed 2 bowel injuries (and one bladder injury) in the first 300 TEP repairs. (www.ncbi.nlm.nih.gov/pubmed/11178763) Therefore bowel and vascular injuries during laparoscopic surgery are real but they are often under reported.

Single incision laparoscopic surgery, where all the instruments are placed in a single port, has the primary aim of preventing vascular and bowel injury through the use of completely blunt trocars as in the case of the SILS™ port. The first case of laparoscopic TEP repair was reported in 2009. Since then there have numerous reports confirming the safety and efficacy of the single-port technique.

The principle author, Dr Hanh Tran, has been performing single incision laparoscopic hernia repair since October 2009. To date, he has performed in excess of 600 cases with excellent results and this was confirmed in a recently completed prospective randomized controlled study comparing single-port vs. multiport laparoscopic inguinal herniorraphy (NCT 01660048) in achieving successful cure of hernias, no complications including wound infection, reduced post-op pain/analgesic requirements, earlier return to work/physical activities, high patient satisfaction and excellent cosmetic results.

However this was achieved at significant additional costs because of the use of the single ports. These costs were not reimbursed by the medical insurance companies. The single-port technique allows for direct insertion of the dissecting instruments into the extraperitoneal space where complete dissection can occur under direct vision as supposed to blind dissection with the balloon dissector just so that two 5mm ports can be inserted during multiport TEP repair.

It is proposed that 51 (or more) patients will be enrolled into the study and this will be compared to the previous 51 patients in the previous RCT with balloon dissection. The single-port TEP inguinal herniorraphy is exactly the same in both procedures except in the telescopic technique the dissection of the extraperitoneal dissection is done under direct vision without the use of the balloon dissector.

The main disadvantage of the single port technique is the relative loss of triangulation and the principle author has shown that this can be overcome with the use of a longer and smaller laparoscope (of which Holroyd Private Hospital has bought two specifically for this purpose), different dissecting techniques and with increased experience. Therefore, if a surgeon is not experienced with this technique the operation and its success can be compromised by inadequate dissection. The author (who has performed over 2500 TEP repairs over the past 13 years) believes that the learning curve for single-port TEP hernia repair for a highly experienced TEP surgeon is around 25-50 ie after this number the operation time will approach that of the standard three ports TEP repair and this has been shown in our recently completed RCT. He has performed in excess of 600 Single-port Laparoscopic hernia repairs since October 2009. Therefore the success of the operation for patients in either arm of the study will not be compromised by lack of experience.

The follow up of these patients will be no different to those followed up under the protocol of the Sydney Hernia Specialists/Clinic. This is a standard follow up and is consistent with normal clinical practice.

In summary, the goals are simple. (i) To perform single-port laparoscopic TEP inguinal herniorraphy with telescopic extraperitoneal dissection; (ii) To assess the efficacy of the newer telescopic dissection technique in a rigorous scientific manner; (iii) To report any unexpected problems or complications; (iv) To follow up patients treated laparoscopically to ensure that the single-port technique with balloon dissection or telescopic dissection have as good results as or better in terms of cure of hernia (absence of recurrence of the hernia) and less complications and better cosmetic results as that which is achieved when the traditional 3-ports technique is used and; (v) to assess the outcomes of patients undergoing telescopic dissection vs. balloon dissection.

ELIGIBILITY:
Inclusion Criteria:

- all patients referred with inguinal/femoral hernias

Exclusion Criteria:

* • workers Compensation cases

  * previous extraperitoneal intervention
  * unfit for a general anaesthetic
  * strangulated hernias

Ages: 16 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients referred with inguinal/femoral hernias from February 2013 will be enrolled into the study
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Post-op pain | measured on day 1 and day 7
  Post-op pain measured on day 1 and 7 using the visual analogue score of 0 to 10

SECONDARY OUTCOMES:
• Conversion to multiport or open operation | up to one year
  This refers to whether any single port procedure needs to be converted to multiports or open procedure. This is quite a normal process as a proportion of multiport procedures are converted to open procedures for safety reasons.
• Length of hospital stay | up to one year
  This assess how long patient stays in hospital whether it is a day procedure or whether they need to stay in hospital overnight or longer
operation time | participants will be followed for the duration of hospital stay, an expected average of 1 day
  this is measured from initial skin incision to complete wound closure
Analgesic requirements | up to one week
  This assesses how many painkiller tablets (Dextropropoxyphene) patients ingest in the first week after operation
return to work or normal physical activities | up to one year
  This assesses how soon patients return to work or normal physical activities
Quality of life health scores | up to 1 year
  SF36 forms are completed before operation, 6 weeks and 1 year after operation
Cosmetic scar score | 1 year
  Scar length will be measured at 6 weeks postop and patients will be asked to assess satisfaction of their own scars 6 weeks and 1 year after surgery
Recurrence of hernia | 1 year
  Patients will be assessed at 1 week, 6 weeks and one year to detect presence of recurrence of hernia
post-operative complications including urinary retention, wound infection, seroma formation, chronic pain, testicular atrophy | 1 year
  Patients will be seen at 1 week, 6 weeks to assess for any peri-operative complications associated with hernia surgery as enumerated above
cost analysis of the ports used | up to one year
  Cost savings arising from telescopic dissection will be assessed using data provided by the Hospital Finance Department regarding the costs of the single ports

CONTACTS AND LOCATIONS:
Overall Officials: Wayne J Hawthorne, MD, Study Chair — The Unviversity of Sydney
Locations (2):
- Australia (2):
  - Holroyd Private Hospital, Guildford, New South Wales
  - St Luke's Hospital, Potts Point, New South Wales

REFERENCES:
- [Result] Tran H. Safety and efficacy of single incision laparoscopic surgery for total extraperitoneal inguinal hernia repair. JSLS. 2011 Jan-Mar;15(1):47-52. doi: 10.4293/108680811X13022985131174. PMID 21902942
- [Result] Tran H. Robotic single-port hernia surgery. JSLS. 2011 Jul-Sep;15(3):309-14. doi: 10.4293/108680811X13125733356198. PMID 21985715
- [Result] Tran H. Safety and efficacy of laparoendoscopic single-site surgery for abdominal wall hernias. JSLS. 2012 Apr-Jun;16(2):242-9. doi: 10.4293/108680812x13427982376301. PMID 23477172
- [Derived] Tran H, Tran K, Turingan I, Zajkowska M, Lam V, Hawthorne W. Single-incision laparoscopic inguinal herniorraphy with telescopic extraperitoneal dissection: technical aspects and potential benefits. Hernia. 2015 Jun;19(3):407-16. doi: 10.1007/s10029-015-1349-6. Epub 2015 Feb 3. PMID 25644488
- See also: Sydney Hernia Specialists Clinic — http://www.herniaspecialists.com.au